CLINICAL TRIAL: NCT05740982
Title: A Phase 2 Randomized, Open-Label, Multisite Trial to Inform Public Health Strategies Involving the Use of MVA-BN Vaccine for Mpox
Brief Title: A Phase 2 Randomized Multisite Trial to Inform Public Health Strategies Involving the Use of MVA-BN Vaccine for Mpox
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-0020B
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03-04

CONDITIONS: Monkeypox
Keywords: Adolescent; Adults; Humoral Immune Response; JYNNEOS; Monkeypox; Mpox; MVA-BN; Non-Inferiority Testing; Non-Randomized; Open-label; Pediatric; Phase 2; Public Health; Vaccine; Vaccinia Naive
MeSH Terms: conditions — Mpox, Monkeypox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4 (Active Comparator): 0.5 mL of 1 x 10^8 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered subcutaneously on adults ages 18-50 years on Days 1 and 29. N=135
  Interventions: Biological: JYNNEOS
- 5 (Experimental): 0.5 mL of 1 x 10^8 (50% Tissue Culture Infectious Dose (TCID50) JYNNEOS (Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN)) administered subcutaneously on adolescents ages 12-17 years on Days 1 and 29. N=315
  Interventions: Biological: JYNNEOS

INTERVENTIONS:
Biological: JYNNEOS — JYNNEOS is FDA-approved and licensed as a smallpox and monkeypox vaccine in the United States. JYNNEOS is a live vaccine produced from the strain Modified Vaccinia Ankara-Bavarian Nordic (MVA-BN), an attenuated, non-replicating orthopoxvirus.

SUMMARY:
This study is a Phase 2 open-label, non-placebo controlled, multi-site clinical trial that will evaluate the standard SC regimen in adolescents ages 12 through 17 years, inclusive, and compared to the standard subcutaneous regimen in adults ages 18 to 50, inclusive. Approximately 135 healthy, vaccinia-naïve adults will be enrolled in a comparator arm (Arm 4) and will be given the standard, licensed regimen of 1x10^8 TCID50 MVA-BN administered SC on Day 1 and 29. These adults (Arm 4) will be combined with the 76 healthy, vaccinia-naïve adults that received the standard SC regimen in Stage 1 (Arm 3). Together, this will be the comparator group for non-inferiority testing for the primary endpoint. Approximately 315 healthy, vaccinia-naïve adolescents will be enrolled and given 1x10^8 TCID50 MVA-BN administered SC on Days 1 and 29 (Arm 5). The study will have a set target enrollment of at least 25% adolescents ages 12 to 14 years, inclusive, to ensure that adequate numbers of younger adolescents are enrolled.

The primary objectives are 1.) to determine if peak (Day 43) humoral immune responses in adolescents ages 12 to 17 years following administration of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC are non-inferior to the response in adults ages 18 to 50 years who received the licensed 2-dose SC regimen of 1 x 10^8 TCID50 MVA-BN ; and 2.) to describe safety of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC in adolescents ages 12 to 17 years.

DETAILED DESCRIPTION:
This study is a Phase 2 open-label, non-placebo controlled, multi-site clinical trial that will evaluate to inform public health decisions regarding the use of JYNNEOS for monkey pox prevention and mitigation of outbreaks. In stage 2 of the study, the standard subcutaneous (SC) regimen in adolescents ages 12 through 17 years, inclusive, and compared to the standard SC regimen in adults ages 18 to 50, inclusive. Approximately 135 healthy, vaccinia-naïve adults will be enrolled in a comparator arm (Arm 4) and will be given the standard, licensed regimen of 1x10^8 TCID50 MVA-BN administered SC on Day 1 and 29. These adults (Arm 4) will be combined with the 76 healthy, vaccinia-naïve adults that received the standard SC regimen in Stage 1 (Arm 3). Together, this will be the comparator group for non-inferiority testing for the primary endpoint. Approximately 315 healthy, vaccinia-naïve adolescents will be enrolled and given 1x10^8 TCID50 MVA-BN administered SC on Days 1 and 29 (Arm 5). The study will have a set target enrollment of at least 25% adolescents ages 12 to 14 years, inclusive, to ensure that adequate numbers of younger adolescents are enrolled.

The primary objectives are 1.) to determine if peak (Day 43) humoral immune responses in adolescents ages 12 to 17 years following administration of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC are non-inferior to the response in adults ages 18 to 50 years who received the licensed 2-dose SC regimen of 1 x 108 TCID50 MVA-BN; and 2.) to describe safety of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC in adolescents ages 12 to 17 years. The secondary objectives are 1) to evaluate humoral immune responses at baseline, prior to the second vaccination, and following receipt of the 2-dose SC regimen of 1 x 10^8 TCID50 MVA-BN in adolescents compared to adults on each study day; 2) to evaluate the kinetics of the humoral immune responses to the 2-dose SC regimen of 1 x 10^8 TCID50 MVA-BN in adolescents and adults through Day 365 after the second dose is administered; 3.) to compare relative safety and reactogenicity between adolescent and adult study arms; and 4.) to evaluate seroconversion between adolescent and adult study arms.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 18 - 50 years of age inclusive at the time of consent; OR Adolescent ages 12 to 17 years inclusive at the time of consent.
2. Adult participant is able to read the written informed consent, states willingness to comply with all study procedures and is anticipated to be available for all study visits; OR Parent(s)/Legal Authorized Representative (LAR)(s) of the participating adolescent is able to read and provides written informed permission and participating adolescent provides assent as appropriate for age or development and approved by IRB. Adolescent states willingness to comply with all study procedures and is anticipated to be available for all study visits.
3. . Adult participant is able to understand and agrees to adhere to Lifestyle Considerations during the study; OR Parent(s)/LAR(s) of the participating adolescent is able to understand and states willingness to comply with Lifestyle Considerations.
4. Females of reproductive potential who have sexual intercourse with males must agree to use highly effective contraception for at least 1 month prior to signing ICF and through Day 57.

   NOTE: See MOP for definitions and list of acceptable and highly effective methods of contraception
5. In good general health as evidenced by medical history, physical examination, and clinical judgement of the investigator to be in stable state of health.

   NOTE: Participants with pre-existing stable chronic medical conditions defined as conditions not requiring significant change in therapy or hospitalization for worsening disease in the 4 weeks prior to enrollment can be included at the discretion of the investigator. This includes stable, well-controlled HIV positive individuals.
6. Individuals with HIV must be on suppressive ART for at least 6 months, report a CD4 count of greater than 350 cells/µL and no AIDS-defining illness in the last year.

Exclusion Criteria:

1. Ever received a licensed or an investigational smallpox or monkeypox vaccine.

   *This includes Dryvax, Acam2000, LC 16 m8, MVA-based vaccine candidate or licensed vaccines, and Jynneos, Imvamune or Imvanex)
2. Any history of monkeypox, cowpox, or vaccinia infection.
3. Close contact of anyone known to have monkeypox in the 3 weeks prior to signing ICF
4. Immunocompromised as determined by the investigator
5. Recent or current use of any immunosuppressing medications in the 4 weeks prior to signing ICF.

   **Topical, ophthalmic, inhaled, intranasal and intraarticular corticosteroids are acceptable, but receipt of >/=20 mg/day of prednisone or equivalent for >/=14 consecutive days in the 4 weeks prior to signing ICF is exclusionary.
6. Pregnant or breast feeding.
7. Received or plans to receive a live vaccine or any COVID-19 vaccine in the 4 weeks before or after each study vaccination.
8. Received or plans to receive any other vaccine in the one week before or after each study vaccination.
9. Received experimental therapeutic agent or vaccine in the 3 months prior to signing ICF.
10. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products.

    ***This includes individuals with history of severe allergic reaction to gentamicin, ciprofloxacin, chicken or egg protein.
11. Has tattoos, scars, or other marks which would, in the opinion of the investigator, interfere with assessment of the vaccination site.
12. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.

    ****This includes acute, subacute, intermittent, or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.
13. Adolescent or adult participant has a history of myocarditis/pericarditis or a history of structural congenital heart defect/cardiac dysrhythmia that, in the opinion of the investigator, poses increased risk to the participant.
14. Adolescent or adult participant has a history of COVID-19 (with positive test for SARS-CoV-2) in the 4 weeks prior to receipt of the first study vaccination.

Note: This includes positive rapid antigen test, polymerase chain reaction (PCR) assay, or other nucleic acid amplification (NAAT) test including those performed by the participant at home.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Events of Special Interest (AESI) in adolescents | Day 1 through Day 210
  Frequency and description of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC in adolescents ages 12 to 17 years.
Occurrence of Medically Attended Adverse Events (MAAE) in adolescents | Day 1 through Day 210
  Frequency and description of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC
Occurrence of Serious Adverse Events (SAEs) in adolescents | Day 1 through Day 394
  Frequency and relatedness of serious Adverse Events (SAE) of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC in for the duration of the study.
Occurrence of solicited Adverse Events (AE) in adolescents | Day 1 through Day 36
  Frequency and severity of solicited systemic and local Adverse Events for 7 days after each vaccination of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC in adolescents ages 12 to 17 years.
Occurrence of unsolicited Adverse Events (AE) in adolescents | Day 1 through Day 57
  Frequency severity, and relatedness of unsolicited Adverse Events after each vaccination of a 2-dose 1 x 10^8 TCID50 MVA-BN regimen administered SC in for adolescents ages 12 to 17 years.
Occurrence of withdrawals and discontinuations of vaccination in adolescents | Day 1 through Day 394
  Frequency of occurrence within adolescents ages 12 to 17 years
Vaccinia virus specific plaque reduction neutralizing antibody (PRNT) Geometric Mean Titers (GMT) | Day 43
  To determine if peak humoral immune responses in adolescents ages 12 to 17 years are non-inferior to adults after receipt of a 2-dose SC regimen of 1 x 10^8 TCID50 MVA-BN.

SECONDARY OUTCOMES:
Frequency of withdrawals or discontinuation of vaccination | Day 1 through Day 394
Occurrence of Adverse Events of Special Interest (AESI) | Day 1 through day 210
  Frequency and description in study arms 1-5
Occurrence of Medically Attended Events (MAAE) | Day 1 through Day 210
  Frequency, description and relatedness in study arms 1-5
Occurrence of Serious Adverse Events (SAE) | Day 1 through Day 394
  Frequency and relatedness in study arms 1-5
Occurrence of solicited Adverse Events (AE) for 7 days after each vaccination | Day 1 through Day 36
  Frequency, severity, and relatedness of solicited systemic and local Adverse Events for 7 days after each vaccination in study arms 1-5.
Occurrence of unsolicited Adverse Events (AE) | Day 1 through Day 57
  Frequency, severity, and relatedness of unsolicited Adverse Events for 28 days after each vaccination; in study arms 1-5
Vaccinia virus specific plaque reduction neutralizing antibody (PRNT) Geometric Mean Titers (GMT) | Day 1 through Day 394
  For adolescents ages 12 to 17 years compared to adults at baseline, prior to the second vaccination, and following receipt of the 2-dose SC regimen of 1 x 10^8 TCID50 MVA-BN.
Vaccinia virus specific plaque reduction neutralizing antibody (PRNT) Geometric Mean Titers (GMT) | Day 29 through Day 394
  Seroconversion in adolescent study arms 1-5
Vaccinia virus specific plaque reduction neutralizing antibody (PRNT) half-life (t ½) | Day 1 through Day 394
  For adolescents ages 12 to 17 years compared to adults following receipt of the 2-dose SC regimen of 1 x 10^8 TCID50 MVA-BN.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - Children's of Alabama Child Health Research Unit (CHRU), Birmingham, Alabama
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - NIH Clinical Research Center, Investigational Drug Management and Research Section, Bethesda, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC University Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Kaiser Permanente Washington Health Research Institute, Seattle, Washington
- Ponce Medical School Foundation Inc., CAIMED Center, Ponce, Puerto Rico

REFERENCES:
- See also: MPox Vaccination Study Survey for adolescent participants interested in enrolling at the University of Rochester Medical Center — http://redcap.urmc.rochester.edu/redcap/surveys/?s=JMH3HYMFDR8NC4TN&ch=nGKWR220ERw3u8y5cf

DOCUMENTS (3):
  • Study Protocol (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/82/NCT05740982/Prot_001.pdf
  • Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT05740982/SAP_002.pdf
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT05740982/ICF_000.pdf